CLINICAL TRIAL: NCT05286281
Title: A PHASE 1, OPEN-LABEL, SINGLE-PERIOD, NON-RANDOMIZED STUDY TO EVALUATE THE PHARMACOKINETICS, EXCRETION, MASS BALANCE AND METABOLISM OF [14C]PF-07265803 ADMINISTERED ORALLY TO HEALTHY ADULT MALE PARTICIPANTS
Brief Title: A Study To Evaluate The Pharmacokinetics, Excretion, Mass Balance and Metabolism of PF-07265803
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C4411010
Record Dates: First submitted 2022-02-14; First posted 2022-03-18 (Actual); Results first posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Healthy
Keywords: LMNA-related DCM; Cardiomyopathy; Lamin Type A; Heart failure; ARRY-371797
MeSH Terms: conditions — Cardiomyopathies; Limb-girdle muscular dystrophy, type 1B; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-07265803 (Experimental): PF-07265803 is a p38 inhibitor formulated for oral delivery.
  Interventions: Drug: PF-07265803

INTERVENTIONS:
Drug: PF-07265803 — PF-07265803 is a p38 inhibitor formulated for oral delivery.

SUMMARY:
The purpose of this study is to assess the pharmacokinetics, excretion, mass balance and metabolism of PF-07265803 (formerly known as ARRY-371797) in approximately 6 healthy adult male participants.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be male and ≥18 years of age at the time of signing the informed consent.
2. Male participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and electrocardiogram (ECG) monitoring.
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests , lifestyle considerations , and other study procedures.
4. Body Mass Index of 18.0 to 32 kg/m2; and a total body weight >50 kg (110 lb).
5. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy, gastric bypass, duodenotomy, colectomy, history of inflammatory bowel disease).
3. History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, or HCVAb. Hepatitis B vaccination is allowed.
4. Participants with a history of irregular bowel movements; e.g., less than 1 bowel movement per day, regular episodes of diarrhea or constipation, irritable bowel syndrome (IBS) or lactose intolerance.
5. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions or situations related to COVID-19 pandemic (eg. Contact with positive case)] that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
6. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study intervention with the exception of moderate/potent CYP3A inducers which are prohibited within 14 days plus 5 half-lives prior to the first dose of study intervention.
7. Current use of any prohibited concomitant medication(s) or those unwilling/unable to use a permitted concomitant medication(s).
8. Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer).
9. A positive urine drug test.
10. Screening and baseline supine blood pressure (BP) >140 mm Hg (systolic) or >90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is >140 mm Hg (systolic) or >90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
11. Screening and baseline standard 12 lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline QTcF interval >450 msec, atrial fibrillation, complete left bundle branch block (LBBB), signs of an acute or indeterminate age myocardial infarction, ST T interval changes suggestive of myocardial ischemia, second or third degree AV block, or serious bradyarrhythmias or tachyarrhythmias). If the baseline uncorrected QT interval is >450 msec, this interval should be rate corrected using the Fridericia method and the resulting QTcF should be used for decision making and reporting. If QTcF exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTcF or QRS values should be used to determine the participant's eligibility. Computer interpreted ECGs should be overread by a physician experienced in reading ECGs before excluding a participant.
12. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

    * Aspartate aminotransferase (AST) or Alanine Aminotransferase (ALT) level ≥ 1.5 × ULN;
    * Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is≤ ULN.
13. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit or 3 ounces (90 mL) of wine).
14. Positive urine drug screen or cotinine at screening or check-in, and positive urine alcohol at check-in.
15. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
16. History of sensitivity to heparin or heparin induced thrombocytopenia.
17. Unwilling or unable to comply with the criteria in the Lifestyle Considerations of this protocol.
18. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.
19. Subjects with exposure to significant diagnostic or therapeutic radiation (eg,serial x ray, computed tomography scan, barium meal) or current employment in a job requiring radiation exposure monitoring within 12 months prior to check-in.
20. Subjects who have participated in more than 3 radiolabeled drug studies in the last 12 months (previous study to be at least 4 months prior to check-in to the study site where exposures are known to the investigator, or 6 months prior to check-in to the study site for a radiolabeled drug study where exposures are not known to the investigator). The total 12-month exposure from this study and a maximum of 2 other previous radiolabeled studies within 4 to 12 months prior to this study will be within the Code of Federal Regulations (CFR) recommended levels considered safe, per United States (US) Title 21 CFR 361.1.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must be male and ≥18 years of age at the time of signing the ICD.
Enrollment: 6 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Labcorp Clinical Research Unit, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4411010

RESULTS

PARTICIPANT FLOW:
Groups:
- [14C]PF-07265803 400 mg: Participants received a single oral dose of PF-07265803 400 mg (containing 100 μCi 14C) on Day 1. μCi = microcurie.
Period: Overall Study
Arm/Group | [14C]PF-07265803 400 mg
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who received at least 1 dose of study treatment.
Groups:
- [14C]PF-07265803 400 mg: Participants received a single oral dose of PF-07265803 400 mg (containing 100 μCi 14C) on Day 1.
Arm/Group | [14C]PF-07265803 400 mg
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.3 (11.74)
Age, Customized [Number; unit: Participants]
  <18 | 0
  18-25 | 0
  26-35 | 0
  36-45 | 2
  >45 | 4
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 6
  Female | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Recovery of Radioactivity in Urine, Expressed as Percentage of Total Radioactive Dose Administered
Description: Radioactivity excreted in urine was reported as the percentage of the administered radioactivity excreted at each time interval, cumulatively through that interval and the total percent of dose recovered in urine.
Time Frame: Predose, in intervals of 0-6, 6-12, 12-24, 24-48, 48-72, 72-96 hours postdose on Day 1, and each subsequent 24 hours interval up to discharge (maximum 14 days)
Population: Extent of excretion population is defined as all participants who received 1 dose of [14C]PF-07265803 and who had evaluable total radioactivity concentration (urinary and fecal) data and who had no protocol deviations or adverse events (such as vomiting of the dose, diarrhoea or severe constipation) that might have affected the extent of excretion analysis.
Measure: Mean (Standard Deviation); unit: Percentage of total radioactive dose
Arm/Group | [14C]PF-07265803 400 mg
Number analyzed (Participants) | 6
Percentage of total radioactive dose | 13.98 (2.3111)

2. Primary Outcome: Total Recovery of Radioactivity in Feces, Expressed as Percentage of Total Radioactive Dose Administered
Description: Radioactivity excreted in feces was reported as the percentage of the administered radioactivity excreted at each time interval, cumulatively through that interval and the total percent of dose recovered in feces.
Time Frame: Predose, in intervals of each 24 hours post dose on Day 1 up to discharge (maximum 14 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of total radioactive dose
Arm/Group | [14C]PF-07265803 400 mg
Number analyzed (Participants) | 6
Percentage of total radioactive dose | 74.65 (3.0842)

3. Primary Outcome: Total Recovery of Radioactivity in Total Excretion (Urine + Feces), Expressed as Percentage of Total Radioactive Dose Administered
Description: Radioactivity excreted in urine and feces was reported as the percentage of the administered radioactivity excreted at each time interval, cumulatively through that interval and the total percent of dose recovered in urine and feces.
Time Frame: Predose, in intervals of each 24 hours post dose on Day 1 up to discharge (maximum 14 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of total radioactive dose
Arm/Group | [14C]PF-07265803 400 mg
Number analyzed (Participants) | 6
Percentage of total radioactive dose | 88.64 (5.0887)

4. Primary Outcome: Relative Abundance of PF-07265803 and Its Metabolites in Plasma, Expressed as Percentage of Radioactivity
Description: Plasma homogenates were extracted for total radioactivity, and processed samples were analyzed by HPLC with radiochemical detection for quantitation of [14C]PF-07265803-derived components and by HRMS for identification of PF-07265803 and metabolites after a single 400-mg (100 μCi) oral dose of [14C]PF-07265803. Relative abundance of the metabolites of [14C]PF-07265803 in plasma based on [14C] quantitation was reported, expressed as percentage of radioactivity. PF-07265803 and four metabolites identified/characterized in human plasma including PF-07327859, PF-07327890, PF -07327860, and des(dimethylamino)-dioxy-PF-07265803 (m/z 461) were presented below. The plasma analysis was done with a single master pool sample (individual participants pooled based on time and from these a single master pool of all participants in one tube) due to the low amount of radioactivity in the plasma, hence there would be no mean or standard deviation.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24, 36, 48, 72, 96, 120 hours post dose on Day 1
Population: All participants who received 1 dose of [14C]PF-07265803 and who had evaluable total radioactivity concentration (urinary and fecal) data and who had no protocol deviations or adverse events (such as vomiting of the dose, diarrhoea or severe constipation) that might have affected the extent of excretion analysis.
Measure: Number; unit: Percentage of radioactivity
Arm/Group | [14C]PF-07265803 400 mg
Number analyzed (Participants) | 6
Percentage of radioactivity
  PF-07265803 | 8.49
  PF-07327859 | 68.27
  PF-07327890 | 12.73
  PF -07327860 | 2.58
  m/z 461 | 2.58

5. Primary Outcome: Relative Abundance of PF-07265803 and Its Metabolites in Urine, Expressed as Percentage of Radioactivity
Description: Urine homogenates were extracted for total radioactivity, and processed samples were analyzed by HPLC with radiochemical detection for quantitation of [14C]PF-07265803-derived components and by HRMS for identification of PF-07265803 and metabolites after a single 400-mg (100 μCi) oral dose of [14C]PF-07265803. In this outcome measure, relative abundance of the metabolites of [14C]PF-07265803 in urine based on [14C] quantitation was reported, expressed as percentage of radioactivity. PF-07265803 and four metabolites identified/characterized in human urine including PF-07327859, PF-07327890, PF-07327891, and des(dimethylamino)-dioxy-PF-07265803 (m/z 461) were presented below.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of radioactivity
Arm/Group | [14C]PF-07265803 400 mg
Number analyzed (Participants) | 6
Percentage of radioactivity
  PF-07265803 | 6.86 (1.33)
  PF-07327859 | 63.9 (4.89)
  PF-07327890 | 11.9 (2.85)
  PF-07327891 | 0.888 (0.754)
  m/z 461 | 1.61 (0.455)

6. Primary Outcome: Relative Abundance of PF-07265803 and Its Metabolites in Feces, Expressed as Percentage of Radioactivity
Description: Fecal homogenates were extracted for total radioactivity, and processed samples were analyzed by HPLC with radiochemical detection for quantitation of [14C]PF-07265803-derived components and by HRMS for identification of PF-07265803 and metabolites after a single 400-mg (100 μCi) oral dose of [14C]PF-07265803. In this outcome measure, relative abundance of the metabolites of [14C]PF-07265803 in feces based on [14C] quantitation was reported, expressed as percentage of radioactivity. PF-07265803 and four metabolites identified/characterized in human urine including PF-07327859, PF-07327890, PF-07327891, and PF-07327860 were presented below.
Time Frame: Predose, in intervals of each 24 hours post dose on Day 1 up to discharge (maximum 14 days)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of radioactivity
Arm/Group | [14C]PF-07265803 400 mg
Number analyzed (Participants) | 6
Percentage of radioactivity
  PF-07265803 | 1.53 (1.48)
  PF-07327859 | 78.1 (3.53)
  PF-07327890 | 6.79 (1.94)
  PF-07327891 | 6.45 (1.12)
  PF-07327860 | 1.90 (1.46)

7. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 to Time of the Last Quantifiable Concentration (AUClast) of Total Radioactivity of [14C]PF-07265803 in Plasma
Description: AUClast is defined as area under the plasma concentration-time profile from time 0 to time of the last quantifiable concentration (Clast). The determination method of AUClast was linear/log trapezoidal rule.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24, 36, 48, 72, 96, 120 hours post dose on Day 1
Population: All participants treated who had at least one of the 14C parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ngEq (nanogram equivalent)*hr/mL
Arm/Group | [14C]PF-07265803 400 mg
Number analyzed (Participants) | 6
ngEq (nanogram equivalent)*hr/mL | 5345 (34)

8. Secondary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) of Total Radioactivity of [14C]PF-07265803 in Plasma
Description: AUCinf is defined as area under the plasma concentration time profile from time zero extrapolated to infinite time.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24, 36, 48, 72, 96, 120 hours post dose on Day 1
Population: All participants treated who had at least one of the 14C parameters of interest. Only 1 participant contributed data for this parameter of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ngEq*hr/mL
Arm/Group | [14C]PF-07265803 400 mg
Number analyzed (Participants) | 1
ngEq*hr/mL | 6430

9. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Total Radioactivity of [14C]PF-07265803 in Plasma
Description: Cmax is defined as maximum plasma concentration. Cmax was observed directly from data.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24, 36, 48, 72, 96, 120 hours post dose on Day 1
Population: All participants treated who had at least one of the 14C parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ngEq/mL (nanogram-equivalent/milliliter)
Arm/Group | [14C]PF-07265803 400 mg
Number analyzed (Participants) | 6
ngEq/mL (nanogram-equivalent/milliliter) | 1183 (13)

10. Secondary Outcome: Time for Cmax (Tmax) of Total Radioactivity of [14C]PF-07265803 in Plasma
Description: Tmax is defined as time for Cmax. Tmax was observed directly from data as time of first occurrence.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24, 36, 48, 72, 96, 120 hours post dose on Day 1
Population: All participants treated who had at least one of the 14C parameters of interest.
Measure: Median (Full Range); unit: hours
Arm/Group | [14C]PF-07265803 400 mg
Number analyzed (Participants) | 6
hours | 1.000 [0.500 to 3.00]

11. Secondary Outcome: Terminal Elimination Half-life (t1/2) of Total Radioactivity of [14C]PF-07265803 in Plasma
Description: Terminal elimination half-life (t1/2) was the time measured for the plasma concentration to decrease by one half. The determination method of t1/2 was loge(2)/kel, where kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24, 36, 48, 72, 96, 120 hours post dose on Day 1
Population: All participants treated who had at least one of the 14C parameters of interest contributing to the summary statistics for t1/2. Only 1 participant contributed data for this parameter of interest.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | [14C]PF-07265803 400 mg
Number analyzed (Participants) | 1
hours | 3.24

12. Secondary Outcome: AUClast of PF-07265803, PF-07327859, PF-07327860 and PF-07327890 in Plasma
Description: as for outcome 7
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24, 36, 48, 72, 96, 120 hours post dose on Day 1
Population: All participants treated who had at least 1 of the PF- 07265803 (or its known circulating metabolites PF-07327859, PF-07327860, PF-07327890) PK parameters of interest contributing to the summary statistics for AUClast.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL (nanogram*hour per milliliter)
Arm/Group | [14C]PF-07265803 400 mg
Number analyzed (Participants) | 6
ng*hr/mL (nanogram*hour per milliliter)
  PF-07265803 | 313.2 (21)
  PF-07327859 | 3661 (17)
  PF-07327860 | 828.3 (109)
  PF-07327890 | 855.5 (27)

13. Secondary Outcome: AUCinf of PF-07265803, PF-07327859, PF-07327860 and PF-07327890 in Plasma
Description: AUCinf is defined as area under the plasma concentration time profile from time zero extrapolated to infinite time. The determination method of AUCinf was AUClast + (Clast*/ kel), where Clast* was the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis, kel was the terminal phase rate constant.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24, 36, 48, 72, 96, 120 hours post dose on Day 1
Population: All participants treated who had at least 1 of the PF-07265803 (or its known circulating metabolites PF-07327859, PF-07327860, PF-07327890) PK parameters of interest contributing to the summary statistics for AUCinf.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | [14C]PF-07265803 400 mg
Number analyzed (Participants) | 6
ng*hr/mL
  PF-07265803 | 315.1 (21)
  PF-07327859: number analyzed (Participants) | 4
  PF-07327859 | 3451 (16)
  PF-07327860: number analyzed (Participants) | 5
  PF-07327860 | 1018 (110)
  PF-07327890 | 871.7 (27)

14. Secondary Outcome: Apparent Clearance (CL/F) of PF-07265803 in Plasma
Description: CL/F is apparent clearance of PF-07265803 from plasma, for extravascular routes of administration. CL/F was calculated with dose/AUCinf.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24, 36, 48, 72, 96, 120 hours post dose on Day 1
Population: All participants treated who had at least 1 of the PF-07265803 (or its known circulating metabolites PF-07327859, PF-07327860, PF-07327890) PK parameters of interest contributing to the summary statistics for CL/F.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr (liter per hour)
Arm/Group | [14C]PF-07265803 400 mg
Number analyzed (Participants) | 6
L/hr (liter per hour) | 1280 (21)

15. Secondary Outcome: Apparent Volume (Vz/F) of PF-07265803 in Plasma
Description: Vz/F is apparent volume of distribution, estimated from terminal phase, for extravascular dosing. Vz/F was calculated with dose /(AUCinf*kel), where kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24, 36, 48, 72, 96, 120 hours post dose on Day 1
Population: All participants treated who had at least 1 of the PF-07265803 (or its known circulating metabolites PF-07327859, PF-07327860, PF-07327890) PK parameters of interest contributing to the summary statistics for Vz/F.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L (liter)
Arm/Group | [14C]PF-07265803 400 mg
Number analyzed (Participants) | 6
L (liter) | 3158 (29)

16. Secondary Outcome: Cmax of PF-07265803, PF-07327859, PF-07327860 and PF-07327890 in Plasma
Description: Cmax is defined as maximum plasma concentration. Cmax was observed directly from data.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24, 36, 48, 72, 96, 120 hours post dose on Day 1
Population: All participants treated who had at least 1 of the PF-07265803 (or its known circulating metabolites PF-07327859, PF-07327860, PF-07327890) PK parameters of interest contributing to the summary statistics for Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | [14C]PF-07265803 400 mg
Number analyzed (Participants) | 6
ng/mL
  PF-07265803 | 258.6 (11)
  PF-07327859 | 741.2 (16)
  PF-07327860 | 22.38 (58)
  PF-07327890 | 117.3 (30)

17. Secondary Outcome: Tmax of PF-07265803, PF-07327859, PF-07327860 and PF-07327890 in Plasma
Description: Tmax is defined as time for maximum plasma concentration (Cmax). Tmax was observed directly from data as time of first occurrence.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24, 36, 48, 72, 96, 120 hours post dose on Day 1
Population: All participants treated who had at least 1 of the PF-07265803 (or its known circulating metabolites PF-07327859, PF-07327860, PF-07327890) PK parameters of interest contributing to the summary statistics for Tmax.
Measure: Median (Full Range); unit: hr (hour)
Arm/Group | [14C]PF-07265803 400 mg
Number analyzed (Participants) | 6
hr (hour)
  PF-07265803 | 0.5000 [0.500 to 0.500]
  PF-07327859 | 1.000 [1.00 to 3.00]
  PF-07327860 | 24.00 [9.00 to 24.0]
  PF-07327890 | 2.500 [2.00 to 4.00]

18. Secondary Outcome: t1/2 of PF-07265803, PF-07327859, PF-07327860 and PF-07327890 in Plasma
Description: as for outcome 11
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 9, 12, 24, 36, 48, 72, 96, 120 hours post dose on Day 1
Population: All participants treated who had at least 1 of the PF-07265803 (or its known circulating metabolites PF-07327859, PF-07327860, PF-07327890) PK parameters of interest contributing to the summary statistics for t1/2.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | [14C]PF-07265803 400 mg
Number analyzed (Participants) | 6
hr
  PF-07265803 | 1.713 (0.14278)
  PF-07327859: number analyzed (Participants) | 4
  PF-07327859 | 4.985 (1.5148)
  PF-07327860: number analyzed (Participants) | 5
  PF-07327860 | 14.79 (7.3121)
  PF-07327890 | 11.97 (6.5779)

19. Secondary Outcome: Number of Participants With All-Causality and Treatment-Related Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. Treatment-related AE was any untoward medical occurrence attributed to study treatment in a participant who received study treatment. Relatedness to study treatment was assessed by the investigator. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study treatment and up to 35 days that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From the first dose of study treatment up to 35 days
Population: All participants assigned to study treatment and who took at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | [14C]PF-07265803 400 mg
Number analyzed (Participants) | 6
Participants
  Number of Participants with all-causality TEAEs | 0
  Number of Participants with all-causality SAEs | 0
  Number of Participants with treatment-related TEAEs | 0
  Number of Participants with treatment-related SAEs | 0

20. Secondary Outcome: Number of Participants With Laboratory Abnormalities Without Regard to Baseline Abnormality
Description: Laboratory abnormalities included: Hemoglobin (HGB), hematocrit, erythrocytes (ery.) <0.8*lower limit of normal (LLN); ery. mean corpuscular (EMC) volume, EMC HGB, EMC HGB concentration, potassium, chloride, calcium, bicarbonate<0.9*LLN,>1.1*ULN; platelets<0.5*LLN,>1.75*upper limit of normal (ULN); leukocytes, glucose<0.6*LLN,>1.5* ULN; lymphocytes, neutrophils, protein, albumin <0.8*LLN,>1.2*ULN; basophils, eosinophils, monocytes, urate >1.2*ULN; bilirubin (total, direct, indirect)>1.5*ULN; aspartate/alanine aminotransferase, alkaline phosphatase>3.0*ULN; sodium <0.95*LLN,>1.05*ULN; blood urea nitrogen, creatinine >1.3*ULN; Urine: pH<4.5,>8; glucose, ketones, protein, HGB, nitrite, leukocyte esterase>=1. Only those categories in which at least 1 participant had data were reported.
Time Frame: From the first dose of study treatment up to 35 days
Population: All participants assigned to study treatment and who took at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | [14C]PF-07265803 400 mg
Number analyzed (Participants) | 6
Participants
  EMC HGB (pg/cell) <0.9*LLN | 1
  Urinalysis: pH (scalar) >8 | 1

21. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs Values
Description: Vital signs (pulse rate, systolic and diastolic blood pressure) were obtained with participant in the supine position, after having approximately 5 minutes of rest. Clinical significance of vital signs was determined at the investigator's discretion.
Time Frame: From the first dose of study treatment up to 35 days
Population: All participants assigned to study treatment and who took at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | [14C]PF-07265803 400 mg
Number analyzed (Participants) | 6
Participants | 0

22. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Values
Description: Standard 12-lead ECGs utilizing limb leads were collected using an ECG machine that automatically calculated the heart rate and measures PR, QT, and QTc intervals and QRS complex. Clinical significance of vital signs was determined at the investigator's discretion.
Time Frame: From the first dose of study treatment up to 35 days
Population: All participants assigned to study treatment and who took at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | [14C]PF-07265803 400 mg
Number analyzed (Participants) | 6
Participants | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 35 days after the last dose of study treatment on Day 1 (up to 35 days)
Arm/Group | [14C]PF-07265803 400 mg
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/81/NCT05286281/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT05286281/SAP_001.pdf